CLINICAL TRIAL: NCT05384262
Title: A Phase I, Randomized, Single-Blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD0780 Following Single and Multiple Ascending Dose Administration to Healthy Subjects With or Without Elevated LDL-C Levels
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD0780 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7960C00001; 2022-002221-10 (EudraCT Number)
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Dyslipidemia
Keywords: Elevated LDL-C; Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, single-blind (study center staff including the Principal Investigator [PI] to remain blinded during the dosing phase of each cohort), placebo-controlled, Single Ascending Dose (SAD)/MAD, parallel type design in healthy male and/or female subjects, performed at multiple study centers.
Who Masked: Participant
Masking Description: This study will be a randomized, single-blind (study center staff including the PI to remain blinded during the dosing phase of each cohort), placebo-controlled, SAD/MAD, sequential group design study in healthy male and/or female subjects, performed at multiple study centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Cohort 1: Part A1 - AZD0780 dose 1/placebo tablet (Active Comparator): A total of 6 subjects will receive single ascending doses of AZD0780 and 2 will receive placebo.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 2: Part A1 - AZD0780 dose 2/placebo tablet (Active Comparator): A total of 6 subjects will receive single ascending doses of AZD0780 and 2 will receive placebo.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 3: Part A1 - AZD0780 dose 3/placebo tablet (Active Comparator): A total of 6 subjects will receive single ascending doses of AZD0780 and 2 will receive placebo.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 4: Part A1 - AZD0780 dose 4/placebo tablet (Active Comparator): A total of 6 subjects will receive single ascending doses of AZD0780 and 2 will receive placebo.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 5: Part A1 - AZD0780 dose 5/placebo tablet (Active Comparator): A total of 6 subjects will receive single ascending doses of AZD0780 and 2 will receive placebo.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 6: Part B - AZD0780 dose 6/placebo tablet (Active Comparator): A total of 20 subjects will be assigned as 3:1::AZD0780:Placebo to receive multiple ascending doses.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 7: Part B - AZD0780 dose 7/placebo tablet (Active Comparator): A total of 20 subjects will be assigned as 3:1::AZD0780:Placebo to receive multiple ascending doses.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 8: Part B - AZD0780 dose 8/placebo tablet (Active Comparator): A total of 20 subjects will be assigned as 3:1::AZD0780:Placebo to receive multiple ascending doses.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 9: Part B - AZD0780 dose 9/placebo tablet (Active Comparator): A total of 6 subjects will receive single and multiple ascending doses of AZD0780 and 2 will receive placebo.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 10: Part B - AZD0780 dose 10/placebo tablet (Active Comparator): A total of 6 subjects will receive single and multiple ascending doses of AZD0780 and 2 will receive placebo.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 11: Part A2 - AZD0780 dose 11/placebo tablet (Active Comparator): A total of 5 subjects will receive single ascending doses of AZD0780 and placebo.
  Interventions: Drug: AZD0780; Drug: Placebo
- Cohort 12: Part B - AZD0780 dose 1/rosuvastatin dose 12 (Active Comparator): A total of 20 subjects will receive single dose of AZD0780 and rosuvastatin.
  Interventions: Drug: AZD0780; Drug: Rosuvastatin
- Cohort 13: Part B - placebo tablet/rosuvastatin dose 12 (Active Comparator): A total of 20 subjects will receive single dose of placebo and rosuvastatin.
  Interventions: Drug: Placebo; Drug: Rosuvastatin
- Cohort 14: Part B - AZD0780 with placebo tablet/AZD0780 with rosuvastatin dose 12 (Active Comparator): A total of 20 subjects will receive AZD0780 in combination with rosuvastatin or 5 subjects will receive placebo in combination with rosuvastatin.
  Interventions: Drug: AZD0780; Drug: Placebo; Drug: Rosuvastatin

INTERVENTIONS:
Drug: AZD0780 — Subjects will receive AZD0780 orally as a single ascending dose.
  Arms: Cohort 11: Part A2 - AZD0780 dose 11/placebo tablet; Cohort 1: Part A1 - AZD0780 dose 1/placebo tablet; Cohort 2: Part A1 - AZD0780 dose 2/placebo tablet; Cohort 3: Part A1 - AZD0780 dose 3/placebo tablet; Cohort 4: Part A1 - AZD0780 dose 4/placebo tablet; Cohort 5: Part A1 - AZD0780 dose 5/placebo tablet
Drug: AZD0780 — Subjects will receive AZD0780 orally as a multiple ascending dose.
  Arms: Cohort 12: Part B - AZD0780 dose 1/rosuvastatin dose 12; Cohort 14: Part B - AZD0780 with placebo tablet/AZD0780 with rosuvastatin dose 12; Cohort 6: Part B - AZD0780 dose 6/placebo tablet; Cohort 7: Part B - AZD0780 dose 7/placebo tablet; Cohort 8: Part B - AZD0780 dose 8/placebo tablet
Drug: AZD0780 — Subjects will receive AZD0780 orally as a single and multiple ascending dose.
  Arms: Cohort 10: Part B - AZD0780 dose 10/placebo tablet; Cohort 9: Part B - AZD0780 dose 9/placebo tablet
Drug: Placebo — Subjects will receive placebo matching the AZD0780 dose orally as a single ascending dose.
  Arms: Cohort 11: Part A2 - AZD0780 dose 11/placebo tablet; Cohort 1: Part A1 - AZD0780 dose 1/placebo tablet; Cohort 2: Part A1 - AZD0780 dose 2/placebo tablet; Cohort 3: Part A1 - AZD0780 dose 3/placebo tablet; Cohort 4: Part A1 - AZD0780 dose 4/placebo tablet; Cohort 5: Part A1 - AZD0780 dose 5/placebo tablet
Drug: Placebo — Subjects will receive placebo matching the AZD0780 dose orally as a multiple ascending dose.
  Arms: Cohort 13: Part B - placebo tablet/rosuvastatin dose 12; Cohort 14: Part B - AZD0780 with placebo tablet/AZD0780 with rosuvastatin dose 12; Cohort 6: Part B - AZD0780 dose 6/placebo tablet; Cohort 7: Part B - AZD0780 dose 7/placebo tablet; Cohort 8: Part B - AZD0780 dose 8/placebo tablet
Drug: Placebo — Subjects will receive placebo matching the AZD0780 dose orally as a single and multiple ascending dose.
  Arms: Cohort 10: Part B - AZD0780 dose 10/placebo tablet; Cohort 9: Part B - AZD0780 dose 9/placebo tablet
Drug: Rosuvastatin — Subjects will receive rosuvastatin orally.
  Arms: Cohort 12: Part B - AZD0780 dose 1/rosuvastatin dose 12; Cohort 13: Part B - placebo tablet/rosuvastatin dose 12; Cohort 14: Part B - AZD0780 with placebo tablet/AZD0780 with rosuvastatin dose 12

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of AZD0780 following single and multiple dose administration to healthy subjects with or without elevated Low-Density Lipoprotein-Cholesterol (LDL-C) levels.

This study will consist of two parts (Parts A and B).

56 subjects have been planned for Part A and 141 subjects for Part B. Additional subjects may be included for the optional cohorts depending upon emerging data.

DETAILED DESCRIPTION:
This is a Phase I, First In Human (FIH), randomized, single-blind, placebo-controlled, study in healthy male and/or female subjects of non-childbearing potential including healthy subjects of Chinese and Japanese ethnicity performed at multiple centers (up to 4 study centers).

56 subjects have been planned for Part A and 141 subjects for Part B.

* Part A:

  * A Screening Period of maximum 28 days.
  * Admission to study center (Day -1 or Day -2).
  * A Treatment Period (Day 1 to Day 3) with a single dose of AZD0780 or placebo on Day 1. Subjects will be discharged on Day 3.
  * A Follow-up Visit within 5 to 7 days after the Investigational Medicinal Product (IMP) dose for all cohorts.
  * An additional Follow-up Visit within 9 to 11 days after the IMP dose from Cohort 3 onwards.

    (i) Part A1 - Up to 5 dose cohorts of AZD0780 are planned to be investigated. Depending on the findings, up to 4 additional dose cohorts may be added. Within each cohort, 6 subjects will be randomized to receive AZD0780, and 2 subjects randomized to receive placebo. Dosing for each ascending dose cohort will proceed with 2 subjects in a sentinel sub-cohort such that one subject will be randomized to receive AZD0780, and one subject will be randomized to receive placebo.

(ii) Part A2 - The subjects from a chosen cohort in Part A1 will return to the study center no sooner than 9 days after the first dose administration of IMP and will receive AZD0780 or placebo after intake of a high-calorie, high-fat breakfast, to assess the effect of food on the PK of AZD0780.

The subjects will stay at the study center until 48 hours post-dose in both the parts.

• Part B:

* Global Multiple Ascending Dose (MAD) cohort - Up to 3 dose cohorts are planned to be investigated. In each cohort, 20 subjects will participate and receive either AZD0780 or placebo, randomized 3:1 for 28 days dosing. Depending on the findings, 3 additional dose levels may be added in up to 3 additional cohorts (up to 20 subjects per cohort).
* Japanese Single and Multiple Ascending Dose (JSMAD) cohorts - Two cohorts are planned. One cohort of 8 Japanese subjects will receive a medium dose level of AZD0780 or placebo randomized 3:1 for 9 days dosing (subjects will receive a single dose of IMP on Day 1 followed by daily dosing on Days 8 to 15 [there is no dose on Days 2 to 7]). The second cohort of 8 Japanese subjects will receive a higher dose level of AZD0780 or placebo.
* Rosuvastatin global MAD cohorts - Two cohorts are planned. Up to 40 subjects in the first cohort will receive either AZD0780 in combination with rosuvastatin or placebo in combination with rosuvastatin, randomized 1:1 to 1 of the 2 treatment arms with 20 subjects per arm. Up to 25 subjects will participate in the second cohort and will be randomized 4:1 to 1 of 2 treatment arms to receive either AZD0780 in combination with rosuvastatin (20 subjects) or placebo in combination with rosuvastatin (5 subjects). Subjects eligible for these cohorts will begin a Screening period of 56 days, a minimum of 21 days run-in period (maximum of up to 28 days), Treatment period of 28 days for each cohort and two Follow-up visits (1 & 2 weeks after last dose of IMP).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures (including the Pre Screening Visit for Part B).
* Healthy male and female subjects (of nonchildbearing potential), aged 18 to 55 years inclusive, with suitable veins for cannulation or repeated venipuncture.
* Females must have a negative pregnancy test at the Screening Visit and on admission to the study center, must not be lactating and must be of non childbearing potential, confirmed at the Screening Visit by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Have a BMI between 18 and 35 kg/m2 inclusive and weigh at least 50 kg and no more than 120 kg inclusive at the Screening Visit and on admission to the study center.
* For Japanese subjects (Part B) and Chinese subjects (Part A):

  1. A subject will be considered Japanese if both parents and all grandparents are Japanese, the subject was born in Japan, and the subject has not lived outside Japan for more than 10 years.
  2. A subject will be considered Chinese if both parents and all grandparents are Chinese, the subject was born in China, and the subject has not lived outside China for more than 10 years.
* For Part B (MAD), at the Screening Visit subjects must have LDL-C ≥ 70 mg/dL but ≤ 190 mg/dL (or ≥ 1.8 mmol/L but ≤ 4.9 mmol/L for London EPCU [Early Phase Clinical Unit]), and triglycerides < 400 mg/dL (or < 10.3 mmol/L for London EPCU).
* For Part B (rosuvastatin global MAD), at the Screening Visit subjects must have LDL-C ≥ 100 mg/dL but < 190 mg/dL (≥ 2.6 mmol/L but ≤ 4.9 mmol/L for London EPCU).

Exclusion Criteria:

* History of any clinically important disease or disorder.
* History or presence of gastrointestinal, hepatic or, renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
* Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) first vaccination within 30 days prior to randomization.
* SARS-CoV-2 second vaccination within 10 days of screening.
* Confirmed Coronavirus disease 2019 (COVID-19) infection during screening and admission, by Polymerase Chain Reaction (PCR) test (in the London EPCU, COVID-19 infection before or during Screening and/or admission will be confirmed by a COVID-19 test. Subjects will undergo COVID-19 testing prior to ICF signing and any subject testing positive will not be screened for the study).
* Any clinically important abnormalities in clinical chemistry, coagulation, hematology, or urinalysis results.
* Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C antibody, and Human immunodeficiency virus (HIV).
* Abnormal vital signs after 10 minutes supine rest at the Screening Visit and on admission to the study center.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12-lead ECG that may interfere with the interpretation of ECG interval measured from the onset of the QRS complex to the end of the T wave (QT) corrected for heart rate (QTc) interval changes including abnormal ST-T-wave morphology at the Screening Visit and/or on admission to the study center.
* Known or suspected history of drug abuse.
* Current smokers or those who have smoked or used nicotine products within the previous 3 months.
* History of alcohol abuse or excessive intake of alcohol.
* Positive screen for drugs of abuse, cotinine (nicotine), or alcohol at Screening and/or admission to the study center.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD0780.
* Excessive intake of caffeine-containing drinks or food.
* Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of any prescribed or nonprescribed medication including antacids, analgesics, herbal remedies, mega-dose vitamins, and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.
* Plasma donation within one month of the Screening Visit or any blood donation/blood loss during the 3 months prior to the Screening Visit.
* Has received another new chemical entity within 30 days or 5 half-lives of the first administration of IMP in this study.
* Subjects who have previously received AZD0780 within 60 days of the first administration of IMP in this study.
* Involvement of any Astra Zeneca or study center employee or their close relatives.
* Any ongoing or recent minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
* Subjects who are vegans or have medical dietary restrictions.
* Subjects who cannot communicate reliably with the investigator.
* Vulnerable subjects.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events | From Screening (≤ 28 days) until Follow-up Visit (5 to 7 days post-dose for all cohorts, and 9 to 11 days post-dose for subjects from Cohort 3 onwards)
  The safety and tolerability of AZD0780 following oral administration of single ascending doses (Part A) and multiple ascending doses (Part B) will be assessed.

SECONDARY OUTCOMES:
Area under plasma concentration time curve from zero to infinity (AUCinf) | SAD cohorts: Day 1-3 until 5-7 days (cohort 1 & 2) & 9-11 days (cohort 3 onwards) post-dose; JSMAD cohorts: Day 1-3,5,8,10,13,15,16 until 7-10 days post-dose; MAD Cohorts: Day 1 to 3,5,8,9,12,15,18,22,25,29 until Days 36, 43 [± 1day]
  The single dose and steady state AUCinf of AZD0780 following oral administration of AZD0780 will be assessed.
Area under plasma concentration time curve from zero to t hours post-dose (AUC[0-t]) | SAD cohorts: Day 1-3 until 5-7 days (cohort 1 & 2) & 9-11 days (cohort 3 onwards) post-dose; JSMAD cohorts: Day 1-3,5,8,10,13,15,16 until 7-10 days post-dose; MAD Cohorts: Day 1 to 3,5,8,9,12,15,18,22,25,29 until Days 36, 43 [± 1day]
  The single dose and steady state AUC(0-t) of AZD0780 following oral administration of AZD0780 will be assessed.
Area under the plasma concentration-curve across the dosing interval (AUCτ) | SAD cohorts: Day 1-3 until 5-7 days (cohort 1 & 2) & 9-11 days (cohort 3 onwards) post-dose; JSMAD cohorts: Day 1-3,5,8,10,13,15,16 until 7-10 days post-dose; MAD Cohorts: Day 1 to 3,5,8,9,12,15,18,22,25,29 until Days 36, 43 [± 1day]
  The single dose and steady state AUCτ of AZD0780 following oral administration of AZD0780 will be assessed.
Maximum observed plasma (peak) drug concentration [Cmax] | SAD cohorts: Day 1-3 until 5-7 days (cohort 1 & 2) & 9-11 days (cohort 3 onwards) post-dose; JSMAD cohorts: Day 1-3,5,8,10,13,15,16 until 7-10 days post-dose; MAD Cohorts: Day 1 to 3,5,8,9,12,15,18,22,25,29 until Days 36, 43 [± 1day]
  The single dose and steady state Cmax of AZD0780 following oral administration of AZD0780 will be assessed.
Amount of unchanged drug excreted into urine from zero to the last quantifiable concentration by interval and cumulatively (Ae[0-last]) | SAD cohorts (Parts A1 & A2): Day 1 to Day 3; JSMAD cohorts (Part B): Day 1 & 15; Global MAD Cohorts Day 1 & 10; Rosuvastatin Global MAD Cohorts (Part B): Day 1 & 8
  The single dose and steady state Ae[0-last] of AZD0780 following oral administration of AZD0780 will be assessed.
Percentage of dose excreted unchanged in urine from zero to the last quantifiable concentration, by interval and cumulatively (fe[0-last]) | SAD cohorts (Parts A1 & A2): Day 1 to Day 3; JSMAD cohorts (Part B): Day 1 & 15; Global MAD Cohorts Day 1 & 10; Rosuvastatin Global MAD Cohorts (Part B): Day 1 & 8
  The single dose and steady state fe[0-last] of AZD0780 following oral administration of AZD0780 will be assessed.
Renal clearance of drug from plasma (CLR) | SAD cohorts (Parts A1 & A2): Day 1 to Day 3; JSMAD cohorts (Part B): Day 1 & 15; Global MAD Cohorts Day 1 & 10; Rosuvastatin Global MAD Cohorts (Part B): Day 1 & 8
  The single dose and steady state CLR of AZD0780 following oral administration of AZD0780 will be assessed.
LDL-C | LDL-C SAD cohorts: Days 1,2,3,5-7,9-11 LDL-C JSMAD cohorts: Days 1,2,3,10,15,16,17;LDL-C Global MAD Cohorts: Days 1,2,3,5,8,12,22, 25,29,36-43;LDL-C Rosuvastatin Global MAD Cohorts:Days -28,-8,-1,1,2,3,5,8,12,15,18,22,29,36-43
  The pharmacodynamics (PD) of AZD0780 by assessment of LDL-C following oral administration of single ascending doses (Part A) and multiple ascending doses (Part B) will be assessed.
Proprotein convertase subtilisin/kexin type 9 (PCSK9) | PCSK9 SAD cohorts: Days 1,2,3;PCSK9 JSMAD cohorts:Days 1,2,3,10,15,16,17,22-25;PCSK9 Global MAD Cohorts:Days 1,8,15,22,29,36-43; PCSK9 Rosuvastatin Global MAD Cohorts:Days 1,8,15,22,29,36-43
  The PD of AZD0780 by assessment of total PCSK9 (and compound stabilized PCSK9 for Part A) following oral administration of single ascending doses (Part A) will be assessed.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Brooklyn, Maryland
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home